CLINICAL TRIAL: NCT01387737
Title: An Open-Label, Multicenter Study to Evaluate the Long-Term Safety, Tolerability and Efficacy of TA-7284 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Long-Term Safety Study of TA-7284 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-7284-06
Record Dates: First submitted 2011-06-28; First posted 2011-07-06 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: TA-7284; JNJ-28431754; Canagliflozin; Sodium Glucose Co-Transporter (SGLT2 inhibitor)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TA-7284-Low (Experimental)
  Interventions: Drug: TA-7284-Low
- TA-7284-High (Experimental)
  Interventions: Drug: TA-7284-High

INTERVENTIONS:
Drug: TA-7284-Low — TA-7284-Low
  Arms: TA-7284-Low
Drug: TA-7284-High — TA-7284-High
  Arms: TA-7284-High

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TA-7284 as monotherapy or combination therapy with other oral anti-hyperglycaemic agent in Japanese patients with Type 2 diabetes mellitus on 52 weeks oral administration.

DETAILED DESCRIPTION:
This is a randomized, 2-arm, parallel group, open-label study to evaluate the safety and efficacy of TA-7284 in Japanese patients with Type 2 diabetes mellitus, who are not optimally controlled on diet and exercise or with oral anti-hyperglycaemic agent. The patients will receive either TA-7284-Low or TA-7284-High orally alone or in combination with oral anit-hyperglycaemic agent for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥20 years old
* Diagnosed with Type 2 diabetes mellitus at least 3 months before screening
* HbA1c of ≥7.0% and ≤10.0% (monotherapy group)
* HbA1c of ≥7.0% and ≤10.5% (combination therapy group)

Exclusion Criteria:

* Type I diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, secondary diabetes mellitus
* Past or current history of severe diabetic complications
* Fasting plasma glucose > 270 mg/dL before treatment start
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients requiring insulin therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1299 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuya Inagaki, M.D., Study Director — Kyoto University, Graduate School of Medicine; Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation
Locations (7):
- Japan (7):
  - Research site, Chugoku
  - Research site, Hokkaido
  - Research site, Kanto
  - Research site, Kinki
  - Research site, Kyushu
  - Research site, Shikoku
  - Research site, Tōhoku

REFERENCES:
- [Derived] Inagaki N, Goda M, Yokota S, Maruyama N, Iijima H. Effects of Baseline Blood Pressure and Low-Density Lipoprotein Cholesterol on Safety and Efficacy of Canagliflozin in Japanese Patients with Type 2 Diabetes Mellitus. Adv Ther. 2015 Nov;32(11):1085-103. doi: 10.1007/s12325-015-0255-8. Epub 2015 Nov 3. PMID 26530268
- [Derived] Inagaki N, Kondo K, Yoshinari T, Kuki H. Efficacy and safety of canagliflozin alone or as add-on to other oral antihyperglycemic drugs in Japanese patients with type 2 diabetes: A 52-week open-label study. J Diabetes Investig. 2015 Mar;6(2):210-8. doi: 10.1111/jdi.12266. Epub 2014 Aug 25. PMID 25802729

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-7284-Low: TA-7284 low dose, once daily for 52 weeks
- TA-7284-High: TA-7284 high dose, once daily for 52 weeks
Period: Overall Study
Arm/Group | TA-7284-Low | TA-7284-High
Started | 584 | 715
Completed | 532 | 641
Not Completed | 52 | 74
Not completed — Adverse Event | 20 | 30
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 3 | 10
Not completed — Withdrawal by Subject | 27 | 31
Not completed — Clearly not eligible for the study | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TA-7284-Low | TA-7284-High | Total
Number analyzed (Participants) | 584 | 715 | 1299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 436 | 520 | 956
  >=65 years | 148 | 195 | 343
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 212 | 375
  Male | 421 | 503 | 924

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Assessed by Adverse Events, Hypoglycemic Events
Time Frame: 54 weeks
Measure: Number; unit: percentage of incidences
Arm/Group | TA-7284-Low | TA-7284-High
Number analyzed (Participants) | 584 | 715
percentage of incidences
  adverse events | 81.8 | 82.8
  hypoglycemia | 14.9 | 13.3

2. Secondary Outcome: Change in HbA1c
Time Frame: Week 52
Reporting Status: Not Posted

3. Secondary Outcome: Change in Fasting Plasma Glucose
Time Frame: Week 52
Reporting Status: Not Posted

4. Secondary Outcome: Change in Body Weight
Time Frame: Week 52
Reporting Status: Not Posted

5. Secondary Outcome: Change in Blood Pressure
Time Frame: Week 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Week 52
Arm/Group | TA-7284-Low | TA-7284-High
Serious Adverse Events (participants affected / at risk) | 30/584 | 32/715
Other Adverse Events (participants affected / at risk) | 371/584 | 464/715
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-7284-Low (N=584) | TA-7284-High (N=715)
Appendicitis (Infections and infestations) | 1 | 2
Chronic sinusitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroiditis subacute (Endocrine disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 3 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Mass (General disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Heat illness (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Suture removal (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TA-7284-Low (N=584) | TA-7284-High (N=715)
Bronchitis (Infections and infestations) | 23 | 29
Cystitis (Infections and infestations) | 15 | 13
Gastroenteritis (Infections and infestations) | 14 | 22
Influenza (Infections and infestations) | 13 | 10
Nasopharyngitis (Infections and infestations) | 176 | 223
Periodontitis (Infections and infestations) | 8 | 17
Pharyngitis (Infections and infestations) | 30 | 37
Vulvovaginal candidiasis (Infections and infestations) | 11 | 17
Hypoglycaemia (Metabolism and nutrition disorders) | 44 | 44
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 54 | 66
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 44 | 59
Constipation (Gastrointestinal disorders) | 28 | 40
Dental caries (Gastrointestinal disorders) | 14 | 24
Diarrhoea (Gastrointestinal disorders) | 12 | 24
Gastritis (Gastrointestinal disorders) | 16 | 13
Eczema (Skin and subcutaneous tissue disorders) | 29 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 15
Pollakiuria (Renal and urinary disorders) | 24 | 29
Thirst (General disorders) | 14 | 17
Blood ketone body increased (Investigations) | 12 | 14
Contusion (Injury, poisoning and procedural complications) | 19 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other